CLINICAL TRIAL: NCT03028038
Title: Evaluation of Efficacy of Injectable Platelet-Rich Plasma (PRP) in Reducing Alveolar Bone Resorption Following Rapid Maxillary Expansion (RME): A Cone Beam Computed Tomography (CBCT) Assessment
Brief Title: Using Platelet Rich Plasma in Reducing Alveolar Bone Resorption During Rapid Maxillary Expansion
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: UDDS-Ortho-04-2016
Record Dates: First submitted 2017-01-18; First posted 2017-01-23 (Estimated); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Bone Resorption
Keywords: Platelet-rich plasma; Rapid maxillary expansion; Buccal bone thickness; Alveolar bone loss; Alveolar bone resorption
MeSH Terms: conditions — Bone Resorption; Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Platelet Rich Plasma (Experimental): Platelet Rich Plasma (PRP) will be injected beneath the buccal periosteal of the first molar and premolar in one mouth side with a split-mouth design before the beginning of Rapid Maxillary Expansion and after 7 days of it.
  Interventions: Drug: Platelet Rich Plasma
- No Platelet Rich Plasma (Experimental): No Platelet Rich Plasma (PRP) will be injected in the other mouth side with a split-mouth design during Rapid Maxillary Expansion.
  Interventions: Drug: No Platelet Rich Plasma

INTERVENTIONS:
Drug: Platelet Rich Plasma — Platelet Rich Plasma (PRP) will be injected beneath the buccal periosteal of the first molar and premolar in one mouth side with a split-mouth design before the beginning of Rapid Maxillary Expansion and after 7 days of it.
  High resolution cone beam computed tomography (CBCT) will be taken before treatment and after 3 months when the Hyrax is removed.
  Other Names: PRP
  Arms: Platelet Rich Plasma
Drug: No Platelet Rich Plasma — No Platelet Rich Plasma (PRP) will be injected in the other mouth side with a split-mouth design during Rapid Maxillary Expansion.
  High resolution cone beam computed tomography (CBCT) will be taken before treatment and after 3 months when the Hyrax is removed.
  Other Names: No PRP
  Arms: No Platelet Rich Plasma

SUMMARY:
The purpose of this study is to determine if the injection of Platelet-rich plasma (PRP) is effective in reducing alveolar bone loss that happens after each rapid maxillary expansion (RME) on the buccal aspect of the posterior teeth.

16 patients with a skeletal maxillary constriction aged between 10-16 years old will get into orthodontic treatment to widen the maxilla using Hyrax appliance.

An amount of patient blood will be withdrawn and centrifuged to get PRP. Then the PRP will be injected in one half of each patient mouth in a split-mouth design, beneath the buccal periosteal of the first molars and first premolars, the halves will be chosen randomly.

High resolution CBCT images will be taken before and after orthodontic treatment to analyze buccal bone thickness and height changes.

DETAILED DESCRIPTION:
Correction of the maxillary transverse discrepancy is essential for treatment of various types of malocclusions. Palatal expansion is the most common method used to improve the transverse dimensions of the maxilla especially Rapid maxillary expansion (RME) . RME is associated with intermittent high force systems which cause lateral flexion of the alveolar processes and buccal displacement of the anchorage teeth . Displacement of these teeth outside the alveolar anatomic limits can damage the periodontium and finally compromising tooth longevity.

Several researchers have studied the incidence of buccal dehiscence and fenestrations after RME , using CBCT Images.

From here It was thought about using a method to eliminate these dangerous side effects. It was found that platelet rich plasma (PRP) has the ability to enhance tissue regeneration, accelerate wound healing and inducing stem cells differentiation through its growth factors (GFs).

This is the first study in the world that will use PRP with orthodontic treatment, because of its benefits and easiness of using in dental clinic.

Study sample, that consists of 16 patients, was calculated using (G-power sample size calculator) depending on the buccal alveolar bone thickness changes, with a study power of 95%.

Sample will be chosen from the patients who are coming to Orthodontic department in the Faculty of dentistry - Damascus university.

Allocation of the sides of intervention (PRP injection) and control sides is made by letting the participants to withdraw a closed envelop from a dark black box. Each envelop in the box contain either (R letter) for the right side or (L letter) for the left side that will be the intervention side for that patient.

After ensuring of the patients compliance with the terms and conditions of this study, the purpose and methods of the study will be explained to the patients using Information Sheet . In case of approval to participate the patients asked to sign the Informed Consent.

Extra & Intra-oral photographs , impressions and clinical examination will be made.

High resolution CBCT will be taken before the beginning of treatment (T0). Hyrax appliance will be applied on the first molars and first premolars and cemented using GIC.

After one day of cementation, 20ml of patients' blood will be withdrawn and centrifuged to get 4 ml of PRP.

The buccal soft tissue will be anesthetized (sub-mucosal) in the intervention side , then the PRP will be injected at the buccal area of the first molar and first premolar in that side using insulin syringe , 2 ml for each tooth mentioned in two points. The first point place is in the middle of the attached gingiva over the mesial root of the first molar and buccal root of the first premolar. The second point is in the mucosal-gingival junction over the same root of each tooth.

Starting of expansion will be done in the same day of injection, twice a day until getting an over correction of 2-3 mm.

After one week, the injection of prp will be repeated in the same way (T1) High resolution CBCT for the maxilla will be taken 3 months after the beginning of treatment (T2).

All measures will be analyzed before and after treatment between two sides. A questionnaire will be given to the patients to study pain level accompanying PRP injection compared to the control side . Pain will be assessed using Visual Analogue Scale (VAS) 1 (No Pain) - 10 (Worst Pain).

A questionnaire will be given to the patients to study their acceptance of new treatment approach with comprehensive orthodontic treatments.

ELIGIBILITY:
Inclusion Criteria:

* 10-16 years old patients
* Complete emergence of first molars and first premolars
* Clinical maxillary transverse deficiency
* Good oral hygiene (Gingival index <1) according to Silness & loe 1964
* ( Plaque index <1)

Exclusion Criteria:

* The presence of a medical situations that affects orthodontic treatment and periodontal health
* The presence of drug therapy affect orthodontic treatment and periodontal health
* Bad oral hygiene (gingival and plaque index >1)
* Patient with physical and psychological limitations
* Metallic restorations or endodontic treatments on the appliance supporting teeth (first molars and first premolars)
* Craniofacial anomalies
* Previous orthodontic treatment
* Patients who did not correctly follow the protocol of activation
* Patients who did not return for control dental appointments
* Patients whose cementation of the appliance failed
* Patients whose dental structures were difficult to visualize on the CBCT scans as a result of artifact

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2018-07-15 (Actual)

PRIMARY OUTCOMES:
Changes in buccal alveolar bone height loss and thickness reduction amount | Evaluation before and after RME. (after 3 months)
  Buccal alveolar bone height loss and thickness reduction amount (The incidence of Dehiscence) as a result of RME (On the intervention compared to non-intervention side) before and after expansion. Assessment will be done using CBCT before treatment (T0) and after 3 months (T2)

SECONDARY OUTCOMES:
Changes in the appliance supporting teeth inclination | Evaluation before and after RME. (after 3 months)
  The changes in the appliance supporting teeth inclination before and after 3 months of orthodontic expansion. Assessment will be done using CBCT before treatment (T0) and after 3 months (T2)
Pain levels | 3 months
  Pain levels accompanying new treatment approach within orthodontic treatment. A questionnaire will be given to the patients on the first day after PRP first injection and after 3 days , 7 days, after 3 months
Patient acceptance | 3 months
  Patient acceptance of the PRP injection during comprehensive orthodontic treatments.A questionnaire will be given to the patients on the first day after Prp first injection and after 3 days , 7 days, after 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Kinda Sultan, MSc, PhD, Study Chair — Damascus University
Locations (1):
- Damascus University, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Agarwal A, Gupta ND. Platelet-rich plasma combined with decalcified freeze-dried bone allograft for the treatment of noncontained human intrabony periodontal defects: a randomized controlled split-mouth study. Int J Periodontics Restorative Dent. 2014 Sep-Oct;34(5):705-11. doi: 10.11607/prd.1766. PMID 25171042
- [Result] Akin M, Baka ZM, Ileri Z, Basciftci FA. Alveolar bone changes after asymmetric rapid maxillary expansion. Angle Orthod. 2015 Sep;85(5):799-805. doi: 10.2319/090214.1. Epub 2014 Dec 5. PMID 25478739
- [Result] Albanese A, Licata ME, Polizzi B, Campisi G. Platelet-rich plasma (PRP) in dental and oral surgery: from the wound healing to bone regeneration. Immun Ageing. 2013 Jun 13;10(1):23. doi: 10.1186/1742-4933-10-23. PMID 23763951
- [Result] Baysal A, Uysal T, Veli I, Ozer T, Karadede I, Hekimoglu S. Evaluation of alveolar bone loss following rapid maxillary expansion using cone-beam computed tomography. Korean J Orthod. 2013 Apr;43(2):83-95. doi: 10.4041/kjod.2013.43.2.83. Epub 2013 Apr 25. PMID 23671833
- [Result] Dhurat R, Sukesh M. Principles and Methods of Preparation of Platelet-Rich Plasma: A Review and Author's Perspective. J Cutan Aesthet Surg. 2014 Oct-Dec;7(4):189-97. doi: 10.4103/0974-2077.150734. PMID 25722595
- [Result] DurmuSlar MC, Alpaslan C, Alpaslan G, Cakir M. Clinical and radiographic evaluation of the efficacy of platelet-rich plasma combined with hydroxyapatite bone graft substitutes in the treatment of intra-bony defects in maxillofacial region. Acta Odontol Scand. 2014 Nov;72(8):948-53. doi: 10.3109/00016357.2014.926023. Epub 2014 Jul 9. PMID 25005628
- [Result] Geramy A, Shahroudi AS. Fixed versus Removable Appliance for Palatal Expansion; A 3D Analysis Using the Finite Element Method. J Dent (Tehran). 2014 Jan;11(1):75-84. Epub 2014 Jan 31. PMID 24910679
- [Result] Gunyuz Toklu M, Germec-Cakan D, Tozlu M. Periodontal, dentoalveolar, and skeletal effects of tooth-borne and tooth-bone-borne expansion appliances. Am J Orthod Dentofacial Orthop. 2015 Jul;148(1):97-109. doi: 10.1016/j.ajodo.2015.02.022. PMID 26124033
- [Result] Lin L, Ahn HW, Kim SJ, Moon SC, Kim SH, Nelson G. Tooth-borne vs bone-borne rapid maxillary expanders in late adolescence. Angle Orthod. 2015 Mar;85(2):253-62. doi: 10.2319/030514-156.1. Epub 2014 Dec 9. PMID 25490552
- [Result] Martinez CE, Gonzalez SA, Palma V, Smith PC. Platelet-Poor and Platelet-Rich Plasma Stimulate Bone Lineage Differentiation in Periodontal Ligament Stem Cells. J Periodontol. 2016 Feb;87(2):e18-26. doi: 10.1902/jop.2015.150360. Epub 2015 Sep 14. PMID 26367495
- [Derived] Alomari EB, Sultan K. Efficacy of injectable platelet-rich plasma in reducing alveolar bone resorption following rapid maxillary expansion: A cone-beam computed tomography assessment in a randomized split-mouth controlled trial. Angle Orthod. 2019 Sep;89(5):705-712. doi: 10.2319/091018-661.1. Epub 2019 Mar 28. PMID 30920874